CLINICAL TRIAL: NCT05238844
Title: A Phase 2a Randomized, Double-blinded, Placebo-controlled, Multi Center, Dose Ranging Study of the Safety and Efficacy of ATI-2173 and Vebicorvir in Combination With Tenofovir Disoproxil Fumarate in Subjects With Chronic Hepatitis B Virus Infection
Brief Title: A Study of Safety and Efficacy of ATI-2173 and Vebicorvir in Combination With Tenofovir Disoproxil Fumarate in Subjects With Chronic Hepatitis B Virus Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor stopped due to partner collaboration ending
Sponsor: Antios Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANTT202
Record Dates: First submitted 2022-01-13; First posted 2022-02-14 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Tenofovir; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ATI-2173 25mg, Vebicorvir 300mg and Tenofovir 300mg (Experimental): Subjects randomized to active arm will receive active 25mg ATI-2173 + active Vebicorvir 300mg + active Tenofovir 300mg
  Interventions: Drug: ATI-2173 25mg; Drug: Vebicorvir 300mg; Drug: Viread 300Mg Tablet
- Tenofovir Disoproxil Fumarate (Active Comparator): Subjects randomized to placebo arm will receive placebo 25mg ATI-2173 + placebo Vebicorvir 300mg + active Tenofovir 300mg
  Interventions: Drug: Viread 300Mg Tablet

INTERVENTIONS:
Drug: ATI-2173 25mg — ATI-2173 is a liver-targeted phosphoramidate prodrug of clevudine designed to enhance anti-HBV activity while decreasing systemic exposure to clevudine. It will be dosed as a capsule by mouth.
  Arms: ATI-2173 25mg, Vebicorvir 300mg and Tenofovir 300mg
Drug: Vebicorvir 300mg — Vebicorvir (formerly ABI-H0731) is an orally administered, potent and selective small molecule inhibitor of the HBV core protein
  Arms: ATI-2173 25mg, Vebicorvir 300mg and Tenofovir 300mg
Drug: Viread 300Mg Tablet — Viread is a nucleotide analogue reverse transcriptase inhibitor used for chronic hepatitis B virus.

SUMMARY:
This is a randomized, double-blinded, placebo-controlled, multi center, dose ranging study of safety and efficacy in volunteers with chronic hepatitis B virus infection. Volunteers will be administered multiple oral doses of ATI-2173 vebicorvir in combination with tenofovir disoproxil fumarate and assessed for safety and efficacy including blood tests to show how the body metabolizes and eliminates the investigational drug as well as how the drug effects the virus infection.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form (ICF)
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. If female, meets one of the following criteria:

   1. Is of childbearing potential and agrees to use an acceptable contraceptive method. Acceptable contraceptive methods include:

      * Abstinence from heterosexual intercourse from the first study drug administration through to at least 6 months after the last dose of the study drug or until completion of the study, whichever is longer
      * Use a non-hormonal intrauterine device, from at least 28 days prior to the first study drug administration through to at least 6 months after the last dose of the study drug or until completion of the study, whichever is longer, with a male condom or a diaphragm/cervical cap plus spermicide from the first study drug administration through to at least 30 days after the last dose of the study drug or until completion of the study, whichever is longer
      * Use of a double-barrier method
      * Male partner vasectomized at least 6 months prior to the first study drug administration Or
   2. Is of non-childbearing potential, defined as surgically sterile (ie, has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation) or is in a postmenopausal state (ie, at least 1 year without menses without an alternative medical condition prior to the first study drug administration and follicle-stimulating hormone [FSH] levels within the normal ranges for postmenopausal state of the clinical site at screening). If the subject engages in sexual relations, a barrier method (male or female condom) should be used to prevent the spread of HBV.
4. If male, meets one of the following criteria:

   a) Is able to procreate and agrees to use one of the accepted contraceptive regimens and not to donate sperm from the first study drug administration to at least 90 days after the last drug administration. An acceptable method of contraception includes one of the following:
   * Abstinence from heterosexual intercourse
   * Male condom with spermicide or male condom with a vaginal spermicide (gel, foam, or suppository) Or c) Is unable to procreate; defined as surgically sterile (ie, has undergone a vasectomy at least 6 months prior to the first study drug administration). If the subject engages in sexual relations, a barrier method (male or female condom) should be used to prevent the spread of HBV.
5. Male or female aged at least 18 years but not older than 70 years
6. Body mass index (BMI) within 18.0 kg/m2 to 35.0 kg/m2, inclusively
7. Light-, non- or ex-smoker (A light smoker is defined as someone using 10.0 nicotine units or less per day for at least 90 days prior to the first study drug administration [refer to APPENDIX 7 for conversions of nicotine usage]. An ex-smoker is defined as someone who completely stopped using nicotine products for at least 6 months prior to the first study drug administration)
8. Serum HBsAg positive at screening and at least 6 months prior to screening.
9. Serum HBeAg positive and HBV DNA ≥ 20,000 IU/mL, or serum HBeAg negative and HBV DNA ≥ 2,000 IU/mL at screening
10. ALT and AST < 5 times the upper limit of normal (ULN) at screening and on the day prior to the first study drug administration (Day -1)

Exclusion Criteria:

1. Female who is lactating at screening
2. Female who is pregnant according to the pregnancy test at screening or prior to the first study drug administration
3. History of significant hypersensitivity to clevudine, tenofovir disoproxil fumarate or any related products (including excipients of ATI-2173, tenofovir disoproxil fumarate, and the placebo) as well as severe hypersensitivity reactions (like angioedema) to any drugs
4. History of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease
5. Presence of clinically significant muscle disorders, myopathies or other forms of liver disease
6. Presence of any clinically significant disease, as captured in the medical history or evidence of findings on the physical examination, vital sign assessment and/or ECG assessment, and that would otherwise exclude subject from eligibility in the context of all other listed inclusion and exclusion criteria, as determined by an Investigator
7. Presence of clinically significant ECG abnormalities at the screening visit, as defined by medical judgment
8. Positive test result for alcohol and/or drugs of abuse at screening or prior to the first drug administration
9. Any history of tuberculosis
10. Active illicit drug use including, but not limited to, cocaine, heroin and methamphetamine (the use of cannabinoids is acceptable)
11. Significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
12. Use of amiodarone in the 28 days prior to the first study drug administration
13. Presence or history of clinically significant gastrointestinal or kidney disease, or surgery that may affect drug bioavailability
14. Cirrhosis of the liver as determined by one of the following:

    * A score greater than F2 for liver fibrosis by FibroScan or FibroSure test within 6 months prior to screening or at the time of screening Or
    * A score greater than F2 on liver biopsy within 12 months prior to screening or at the time of screening
15. History of or known presence of hepatocellular carcinoma
16. Acute infection or any other clinically significant illness within 14 days of Day 1 of the study
17. History of organ transplantation
18. Presence of uncontrolled hypertension
19. Positive screening results to HIV Ag/Ab combo or hepatitis C virus tests
20. Any other clinically significant abnormalities in laboratory test results at screening that would, in the opinion of an Investigator, increase the subject's risk of participation, jeopardize complete participation in the study, or compromise interpretation of study data
21. Intake of an Investigational Product (IP) in the 28 days prior to the first study drug administration
22. Donation of 50 mL or more of blood in the 28 days prior to the first study drug administration
23. Donation of 500 mL or more of blood in the 56 days prior to the first study drug administration
24. Previous approved or investigational treatment for HBV, including nucleoside therapy, other than treatment by tenofovir or interferon alpha. Prior treatment with tenofovir or interferon alpha must have been discontinued at least 6 months prior to Screening.
25. Positive screening results to hepatitis D virus (HDV) tests
26. History of significant hypersensitivity to excipients of vebicorvir or its placebo
27. Current or prior use of prohibited concomitant medications as defined in Section 4.5.1.
28. Participation in the ANTT201 study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
The percentage of subjects who experienced at least 1 treatment-emergent adverse event (TEAE) | Through study completion, an average of 1 year
The percentage of subjects who experienced at least 1 treatment-emergent serious adverse event (TE SAE) | Through study completion, an average of 1 year
The percentage of subjects who experienced a treatment-emergent dose-limiting toxicity (TE DLT) | Through study completion, an average of 1 year
The percentage of subjects who experienced at least 1 treatment-emergent Division of AIDS (DAIDS) Grade 1, 2, 3, 4, or 5 laboratory abnormality | Through study completion, an average of 1 year
The percentage of subjects who discontinued the study drug due to a TEAE | Through study completion, an average of 1 year
Alanine aminotransferase and aspartate aminotransferase levels versus time | Through study completion, an average of 1 year
Time to HBV viral load relapse in HBV-infected subjects as measured by HBV DNA viral load in IU/mL | Through study completion, an average of 1 year, which is 6 months after end of treatment

SECONDARY OUTCOMES:
Baseline-adjusted maximal reduction in HBV DNA viral load (Emax,HBV) through 6 months after end of treatment following ATI-2173 + vebicorvir + TDF or placebo + TDF for 90 days in HBV-infected subjects | Through study completion, an average of 1 year, which is 6 months after end of treatment
TEmax,HBV through 6 months after end of treatment following ATI-2173 + vebicorvir + TDF or placebo + TDF for 90 days in HBV-infected subjects | Through study completion, an average of 1 year, which is 6 months after end of treatment
AUEC(HBV) through 6 months after end of treatment following ATI-2173 + vebicorvir + TDF or placebo + TDF for 90 days in HBV-infected subjects | Through study completion, an average of 1 year, which is 6 months after end of treatment
Proportion of subjects with HBV DNA sustained viral response as measured by HBV DNA viral load at 6 months after end of treatment | Through study completion, an average of 1 year, which is 6 months after end of treatment
Cmax of ATI-2173, clevudine and M1 in plasma | Through study completion, an average of 1 year
Tmax of ATI-2173, clevudine and M1 in plasma | Through study completion, an average of 1 year
Ctrough of ATI-2173, clevudine and M1 in plasma | Through study completion, an average of 1 year
Ctau of ATI-2173, clevudine and M1 in plasma | Through study completion, an average of 1 year
AUC0-24 of ATI-2173, clevudine and M1 in plasma | Through study completion, an average of 1 year
AUCtau of ATI-2173, clevudine and M1 in plasma | Through study completion, an average of 1 year
t1/2 of ATI-2173, clevudine and M1 in plasma | Through study completion, an average of 1 year
RAC(Cmax) of ATI-2173, clevudine and M1 in plasma | Through study completion, an average of 1 year
RAC(AUC) of ATI-2173, clevudine and M1 in plasma | Through study completion, an average of 1 year
Proportion of subjects with HBV SVR12, SVR18, and SVR24months | Through study completion, an average of 1 year, or through 24 months if applicable
Proportion of subjects with on-treatment ALT flares | Through Day 90
Proportion of subjects with off-treatment ALT flares | From Day 90 through end of study, about 6 months
Rate of HBV viral load return to baseline off-treatment | From Day 90 through end of study, about 6 months
Relationship between HBV RNA and HBV Sustained Viral Response at 6 months | Through study completion, an average of 1 year, which is 6 months after treatment
Change from baseline value in HBV RNA at end of treatment and Sustained Viral Response at 6 months | Through study completion, an average of 1 year, 6 months after treatment
Change from baseline in HBsAg over time and Sustained Viral Response at 6 months | Through study completion, an average of 1 year, 6 months after treatment
Change from baseline value in HBcrAg at end of treatment and Sustained Viral Response at 6 months | Through study completion, an average of 1 year, 6 months after treatment
Relationship between HBV DNA Sustained Viral Response and HBsAg | Through study completion, an average of 1 year
Reduction from baseline in HBsAg following ATI-2173 + vebicorvir + TDF or placebo + TDF for 90 days in HBV-infected subjects | Through study completion, an average of 1 year
Reduction from baseline in HBV RNA following ATI-2173 + vebicorvir + TDF or placebo + TDF for 90 days in HBV-infected subjects | Through study completion, an average of 1 year
Reduction from baseline in HBcrAg following ATI-2173 + vebicorvir + TDF or placebo + TDF for 90 days in HBV-infected subjects | Through study completion, an average of 1 year
Cmax of tenofovir in plasma | Through study completion, an average of 1 year
Tmax of tenofovir in plasma | Through study completion, an average of 1 year
Ctrough of tenofovir in plasma | Through study completion, an average of 1 year
Ctau of tenofovir in plasma | Through study completion, an average of 1 year
AUC0-24 of tenofovir in plasma | Through study completion, an average of 1 year
t1/2 of tenofovir in plasma | Through study completion, an average of 1 year
RAC(Cmax) of tenofovir in plasma | Through study completion, an average of 1 year
RAC(AUC) of tenofovir in plasma | Through study completion, an average of 1 year
Cmax of vebicorvir in plasma | Through study completion, an average of 1 year
Tmax of vebicorvir in plasma | Through study completion, an average of 1 year
Ctrough of vebicorvir in plasma | Through study completion, an average of 1 year
Ctau of vebicorvir in plasma | Through study completion, an average of 1 year
AUC0-24 of vebicorvir in plasma | Through study completion, an average of 1 year
t1/2 of vebicorvir in plasma | Through study completion, an average of 1 year
RAC(Cmax) of vebicorvir in plasma | Through study completion, an average of 1 year
RAC(AUC) of vebicorvir in plasma | Through study completion, an average of 1 year
Correlation between individual tie to viral load relapse and Day 90 clevudine, vebicorvir, and tenofovir Cmin and AUC | Through study completion, an average of 1 year
Correlation between SVR6 and Day 90 clevudine, vebicorvir, and tenofovir Cmin and AUC | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- Republican Clinical Hospital "Timofei Mosneaga" Arensia EM Unit, Chisinau, Republic of Moldova, Moldova
- Medical Center of Limited Liability Company "Harmoniya krasy", Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No